CLINICAL TRIAL: NCT01511575
Title: Analysis of MicroRNA Expression in Down Syndrome Acute Myeloid Leukemia and the Transient Myeloproliferative Disorder
Brief Title: Studying Biomarker Expression in Samples From Patients With Down Syndrome and Acute Myeloid Leukemia or Other Transient Myeloproliferative Disorder
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML12B3; COG-AAML12B3 (Other: Children's Oncology Group); AAML12B3 (Other: Children's Oncology Group); NCI-2012-00111 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-01-13; First posted 2012-01-18 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia in remission; childhood acute myeloid leukemia/other myeloid malignancies; childhood acute megakaryocytic leukemia (M7)
MeSH Terms: conditions — Leukemia | interventions — Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood, tissue, and bone marrow from patients with cancer in the laboratory may help doctors learn about changes that occur in RNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies RNA samples from patients with Down syndrome and acute myeloid leukemia or other transient myeloproliferative disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare miRNA expression in distinctive diagnostic groups: transient myeloproliferative disorder (TMD), Down syndrome (DS) acute megakaryocytic leukemia (AMkL), non-DS AMkL, and in remission DS samples (representing germline, non-malignant samples).

OUTLINE: Archived RNA samples are analyzed for mature micro (mi)RNA expression by real-time RT-PCR. Results are then compared with miRNA expression of non-Down syndrome patients with acute megakaryocytic leukemia.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with Down syndrome (DS) diagnosed with acute myeloid leukemia or transient myeloproliferative disorder
* Clinical samples obtained from patients enrolled on the COG AAML0431 and COG AAML08B1

PATIENT CHARACTERISTICS:

* Previously consented to biologic studies

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with Down syndrome (DS) diagnosed with acute myeloid leukemia or transient myeloproliferative disorder.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Gene expression levels between DS AMKL and non-DS AMKL patients

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Taub, MD, Principal Investigator — Children's Hospital of Michigan